CLINICAL TRIAL: NCT01464047
Title: Korean Post-marketing Surveillance for Sprycel®
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA180-370
Record Dates: First submitted 2011-10-10; First posted 2011-11-03 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Leukemia, Myelomonocytic, Chronic; Leukemia-Lymphoma
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with CML or Ph+ ALL

SUMMARY:
The purpose of this post-marketing surveillance is to investigate and confirm the type and incidence of newly identified adverse events and any other factors affecting safety and efficacy of Sprycel® so that the regulatory authority can manage the marketing approval properly.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with Philadelphia chromosome-positive (Ph+) chronic myeloid leukemia (CML) in chronic phase
* Adults with chronic, accelerated, or myeloid or lymphoid blast phase Ph+ CML with resistance or intolerance to prior therapy including Imatinib
* Adults with Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ALL) with resistance or intolerance to prior therapy

Exclusion Criteria:

* According to Warning/Caution in local label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic myeloid leukemia (CML) or Philadelphia chromosome positive acute lymphoblastic leukemia (Ph+ ALL) who were never treated with Sprycel®
Sampling Method: Non-Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2011-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Adverse events occurrence | 30 days after last dose of study drug

SECONDARY OUTCOMES:
Improvement in hematologic response | 4 weeks after registration
  The number and percentage of subjects who satisfy each criterion of hematologic responses (Complete/No response) will be presented as frequency distribution. McNemar test will be conducted to test the change from the baseline value
Improvement in cytogenetic response | 12 weeks after registration
  The number and percentage of subjects who satisfy each criterion of cytogenetic responses (Complete/Partial/Minor/Minimal/No response) will be presented as frequency distribution. McNemar test will be conducted to test the change from the baseline value
Overall efficacy assessment by investigator's discretion | 4 weeks after registration
  Based on demographic factors, treatment factors like medical history and concomitant medication

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Seoul, South Korea

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx